CLINICAL TRIAL: NCT05925595
Title: A Randomized, Parallel Group, Single Blind Clinical Trial Against Active Comparator to Evaluate the Efficacy and Safety of a Medical Device Made of a Vegetal Biological Matrix for the Treatment of Knee Osteoarthritis.
Brief Title: Intra-articular Administration of Med Device Made of Biological Vegetal Matrix for the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bios-Therapy, Physiological Systems for Health S.p.A (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NBM-KOA 05/21
Record Dates: First submitted 2023-06-22; First posted 2023-06-29 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2023-06

CONDITIONS: the Treatment of Knee Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single blinded (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental): Arm: Medical Device Iniettabile Ginocchio
  Interventions: Device: Medical Device Iniettabile Ginocchio
- Comparator Arm (Active Comparator): Arm: Medical Device Jonexa (active comparator medical device from the market )
  Interventions: Device: Medical Device Iniettabile Ginocchio

INTERVENTIONS:
Device: Medical Device Iniettabile Ginocchio — Knee injection of the investigational device( MD Iniettabile Ginocchio) versus active comparator (Jonexa).

SUMMARY:
A pre-market randomized, parallel group, single-blind, clinical study with a Medical Device, made of vegetal material, to evaluate the efficacy and safety of one knee injection of the investigational device versus active comparator (Jonexa). The study population will consist of 150 patients diagnosed with primary knee osteoarthrosis. At present, the study is monocentric competitive.

Treatment period for each patient is 6 months.

DETAILED DESCRIPTION:
150 patients diagnosed with primary knee osteoarthritis will be enrolled by up to 3 centers.

The study includes 7 visits at the site center.

V-1 (eligibility assessment / screening visit):

* Collection of written informed consent
* Physical examination, including measurement of anthropometric parameters and vital signs (height, weight, diastolic / systolic pressure, heart rate)
* Diagnosed with radiologically confirmed primary osteoarthritis of the knee according to American College of Rheumatology criteria (i.e. one or more osteophytes and a measurable joint space on a plain radiograph taken within 3 months prior to screening).
* Blood tests: glycemia, creatinine, complete blood count with formula, ALT, AST, ALP, calcium, potassium, sodium, C reactive protein, total bilirubin. Urinalysis.
* Advice on daily diary writing to collect the number of concomitant medication before V0
* Recording of adverse events and concomitant therapies in the daily diary

V0 (confirmation of possession of selection criteria):

* Physical examination, including measurement of anthropometric parameters and vital signs (height, weight, diastolic / systolic pressure, heart rate)
* Randomization 1:1 to Investigational device or active comparator Jonexa
* Intra-articular administration
* Observation of the patient for 30 minutes post injection
* Compliance with daily diary completion
* Administration of questionnaires: WOMAC Pain and Function, SF-36 and global symptom relief questionnaire (CGI- I).
* Recording of any changes in concomitant therapies and any adverse events.

V1(Day 3): safety visit (3 days after V0)

* Objective examination, including measurement of vital parameters (weight, diastolic/systolic blood pressure, heart rate).
* Safety evaluation and AEs recording and Concomitant Therapies
* Checking the completion of the daily diary.

V2 (V2, week 2 ± 2 days) follow-up visit:

* Objective examination, including measurement of vital parameters (weight, diastolic/systolic blood pressure, heart rate).
* Checking the completion of the daily diary.
* Administration of the global symptom relief questionnaire (CGI- I).
* Administration of the WOMAC Pain questionnaire.
* Recording of adverse events and concomitant therapies.
* Instruction to fill in the daily diary via web app (smart phone) to report the use of all concomitant therapies. If patient is not able to use web app, a paper copy will be given.

V3 (V3, week 4 ± 2 days): follow-up visit:

* Objective examination, including measurement of vital parameters (weight, diastolic/systolic blood pressure, heart rate).
* Checking the completion of the daily diary.
* Administration of the global symptom relief questionnaire (CGI- I).
* Questionnaire administration: WOMAC Pain and Function, SF-36.
* Recording of adverse events and concomitant therapies.
* Instruction to fill in the daily diary via web app (smart phone) to report the use of all concomitant therapies. If patient is not able to use web app, a paper copy will be given.

V4 (V4, week 12 ± 2 days) follow-up visit:

* Physical examination, including measurement of anthropometric parameters and vital signs (height, weight, diastolic / systolic pressure, heart rate)
* Check of daily diary
* Administration of the global symptom relief questionnaire (CGI- I).
* Questionnaire administration: WOMAC Pain and Function, SF-36.
* Recording of adverse events and concomitant therapies.
* Instruction to fill in the daily diary via web app (smart phone) to report the use of all concomitant therapies. If patient is not able to use web app, a paper copy will be given.

V5 (V5, week 24 ± 3 days) end-of-study or premature discontinuation visit:

* Objective examination, including measurement of vital parameters
* Blood tests: blood glucose, creatinine, blood count with formula,AST, ALP, calcemia, potassium, sodium, C-reactive protein, total bilirubin. Urine examination.
* Check of completion of the daily diary.
* Administration of the global symptom relief questionnaire (CGI- I).
* Questionnaire administration: WOMAC Pain and Function, SF-36.
* Recording of adverse events and concomitant therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Patient of both sexes over 40 years of age
3. Diagnosis of primary osteoarthritis of the knee according to the criteria of the American College, radiologically confirmed, i.e., one or more osteophytes and a measurable joint space on a standard radiograph taken within 3 months prior to screening.
4. Score ≥2 in the target knee on a Likert scale at WOMAC pain question 1 (i.e. pain while walking on a flat surface) at the V-1 screening visit (to be confirmed at the V0 baseline visit). The target knee is defined as the knee with osteoarthritis in the case of unilateral pathology or the only one with this criterion in the case of bilateral pathology.
5. Severity grade of arthrosis 2 or 3 according to Kellgren & Lawrence classification.
6. Be willing to maintain stable eating habits and lifestyle throughout the study period

Exclusion Criteria:

1. Intake of analgesics, NSAIDs or opioids within 5 days prior to the start of the run-in (i.e. prior to V-1).
2. Body Mass Index (BMI) ≥ 30 kg/m2 .
3. Pregnant women.
4. Intra-articular visco supplementation in the target knee in the preceding 9 months.
5. Cycle of treatment with systemic corticosteroids or intra-articular corticosteroid injection in any joint in the 3 months prior to screening.
6. Symptomatic arthrosis of the contralateral knee with a score ≥3 on a Likert scale to WOMAC pain question 1 (pain while walking on a flat surface) at V-1 (to be confirmed at V0), or severe symptomatic hip arthrosis.
7. Significant deformity: genu varum, ligament laxity or meniscus instability.
8. Presence of autoimmune diseases (excluding chronic autoimmune thyroiditis) or other chronic inflammatory processes (e.g. rheumatoid arthritis, ongoing infections, gout).
9. Ongoing infections.
10. Established or presumed allergy to hyaluronic acid, echinacea or centella.
11. Patients with malignant neoplasms of any kind, or with a history of malignant neoplasms except for patients with a positive history of a malignant neoplasm that has been surgically removed and has not recurred within five years prior to study participation.
12. Abuse of alcohol, narcotics or psychotropic drugs that can alter the state of vigilance and physical perception.
13. Dementia of any kind or other possible causes of progressive deterioration of the mental soundness, or any psychological or physical disability that reduces the ability to take the treatment under study as intended.
14. Inadequate reliability or presence of conditions that may lead to non- compliance/adherence of the patient to the protocol.
15. Previous participation in a clinical study within the last 30 days.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Change at 2 weeks from baseline in WOMAC Pain | [Time Frame: 14 days]
  To the patient will be asked to answer 5 questions about the pain experienced in the previous 48 hours, during different activities, using a 5-point Likert scale (0 to 4) for each answer. The total score (minimum 0; maximum 20) is given by the sum of the 5 answers given.

SECONDARY OUTCOMES:
Change from baseline in WOMAC function | Time Frame: 14 days
  To the patient will be asked to answer 16 questions about the function in the previous 48 hours, during different activities, using a 5-point Likert scale (0 to 4) for each answer. The total score
Change in WOMAC pain and function at 4, 12, 24 weeks from baseline | Time Frame: baseline, 4, 12, 24 weeks
  To the patient will be asked to answer " WOMAC pain and function" questions about the function in the previous 48 hours, during different activities, using a 5-point Likert scale at 4, 12, 24 weeks from baseline
Change in SF-36 at 4, 12, 24 weeks from baseline | Time Frame: baseline, 4, 12, 24 weeks
  To the patient will be asked to answer " Change in SF-36 "at 4, 12, 24 weeks from baseline
Adequate global relief of symptoms after treatment | Time Frame: 2, 4, 12, 24 weeks
  Adequate global relief of symptoms after treatment, defined by a score of at least 3 on a 7-point Likert scale of weekly relief (Clinical Global Impression - Improvement, (CGI-I) scale):
  In order to assess adequate global relief, patients will be asked at each post-basal visit (from visit V2 onwards) to answer the question "Compared to how you usually felt before taking the study treatment, how would you rate your global symptom relief over the last 7 days?" Possible answers: 1, much improved; 2, improved; 3, slightly improved; 4, unchanged; 5, slightly worsened; 6, worsened; 7, much worsened.

CONTACTS AND LOCATIONS:
Overall Officials: Auro Caraffa, MD, Principal Investigator — Azienda Ospedaliera di Perugia
Locations (1):
- Azienda Ospedaliera di Perugia, Perugia, Perugia, Italy

IPD SHARING:
Plan to Share IPD: No